CLINICAL TRIAL: NCT04072822
Title: A Multicenter, Randomized, Double Blinded, Placebo-controlled Clinical Trial of Anakinra (Plus Zinc) or Prednisone in Patients With Severe Alcoholic Hepatitis by the AlcHepNet Consortium
Brief Title: Trial of Anakinra (Plus Zinc) or Prednisone in Patients With Severe Alcoholic Hepatitis
Acronym: AlcHepNet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Samer Gawrieh, Clinical-Director, Alcoholic Hepatitis Network Data Coordinating Center and Associate Professor of Clinical Medicine Division of Gastroenterology and Hepatology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AlcHepNet-02
Record Dates: First submitted 2019-08-09; First posted 2019-08-28 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Interleukin 1 Receptor Antagonist Protein; Zinc; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prednisone (Active Comparator): Standard of care plus prednisone 40 mg orally once daily on Days 1-30 and matching placebos for Anakinra (1 syringe s.c. once daily on Days 1-14), and zinc (matched pill once daily on Days 1-90).
  Interventions: Drug: Prednisone; Drug: Placebos
- Anakinra and Zinc (Active Comparator): Standard of care plus Anakinra (100 mg s.c.) once daily on Days 1-14 zinc sulfate 220 mg once daily on Days 1-90, and placebo for prednisone (matched pill once daily on Days 1-30).
  Interventions: Drug: Anakinra and Zinc; Drug: Placebos

INTERVENTIONS:
Drug: Anakinra and Zinc — Anakinra is indicated for reduction in signs and symptoms and slowing the progression of structural damage in moderately to severely active rheumatoid arthritis. It has been previously studied in AH. Zinc is a nutritional supplement. Zinc supplementation reverses the clinical signs of zinc deficiency in participants with alcoholic liver disease.
  Arms: Anakinra and Zinc
Drug: Prednisone — Prednisone is indicated for numerous conditions including inflammatory disease. Corticosteroids, such as prednisolone, are considered standard of care in alcoholic liver disease.
  Arms: Prednisone
Drug: Placebos — Matching placebo

SUMMARY:
This multicenter, randomized, double blinded, placebo-controlled clinical trial is focused on novel treatments for severe alcoholic hepatitis (AH), a life-threatening stage of alcoholic liver injury that has a short-term mortality rate much higher than that of other liver diseases.

The primary objective of the study is to determine the clinical efficacy and safety of Anakinra (plus zinc) compared to the current standard medical treatment consisting of prednisone in participants with clinically severe AH. Key secondary objectives broadly are as follows: (a) to evaluate the use of biomarkers to assess disease severity and treatment response; and (b) to develop novel endpoints to overcome the limitations of current assessment strategies for severe AH.

ELIGIBILITY:
Inclusion Criteria

1. AH, as defined by the NIAAA pan-consortia for AH:

   1. Onset of jaundice (defined as serum total bilirubin >3 mg/dL) within the prior 8 weeks to screening visit
   2. Regular consumption of alcohol with an intake of > 40 gm daily or >280gm weekly on average for women and > 60 gm daily or >420gm weekly on average for men for 6 months or more, with less than 8 weeks of abstinence before onset of jaundice
   3. AST > 50 IU/l
   4. AST:ALT > 1.5 and both values < 400 IU/l
   5. and/or histological evidence of AH*
2. MELD 20-35 on day of randomization.
3. Ages >21

   * In patients with possible AH or AH with confounding factors such as possible ischemic hepatitis, possible DILI, uncertain history of alcohol use (e.g., patient denies excessive alcohol use), and atypical/abnormal laboratory tests (e.g., AST < 50 IU/L or > 400 IU/L, AST/ALT ratio < 1.5), antinuclear antibody > 1:160 or SMA > 1:80, a standard of care liver biopsy may be performed during current hospital admission to confirm AH and exclude competing etiologies

Exclusion Criteria

1. MELD SCORE <20 or > 35
2. Active sepsis (positive blood or ascitic cultures) with Systemic Inflammatory Response Syndrome (SIRS) or hemodynamic compromise requiring intravenous pressors to maintain tissue perfusion
3. Pneumonia as evidenced by radiological exam
4. Multi-organ failure
5. Renal failure defined by GFR <35 mL/min by CKD-EPI.
6. Clinically active C. diff infection
7. History of imaging of the liver (ultrasound, computerized tomography or magnetic resonance) showing other causes of jaundice
8. History of other liver diseases including hepatitis B (positive HBsAg or HBV DNA), hepatitis C (positive HCV RNA), autoimmune hepatitis, Wilson disease, genetic \hemochromatosis, alpha1-antitrypsin deficiency or strong suspicion of Drug Induced Liver Injury (DILI). Previously treated hepatitis C that was cured (sustained virological response with negative RNA ≥24 weeks following treatment) is not an exclusion.
9. History of HIV infection (positive HIV RNA or on treatment for HIV infection)
10. History or presence of cancer (including hepatocellular carcinoma) other than non- melanoma skin cancer
11. History of other significant medical problems such as autoimmune diseases, severe asthma, psoriasis, Inflammatory Bowel Disease (IBD), etc. that might require immunosuppressive treatments
12. Pregnancy or breastfeeding
13. Prior exposure to experimental therapies in last 3 months
14. Prior exposure to systemic corticosteroid (glucocorticoid) or immunosuppressive therapy for more than 4 days within previous 30 days
15. Need for inotropic pressor support to maintain perfusion to critical organs within prior 48 hours before randomization and initiation of experimental treatment
16. Clinically significant pancreatitis- abdominal pain, elevated lipase (> 3 X ULN) and at least edema of pancreas with fat-stranding on CT scan
17. Total WBC count > 30,000/mm3
18. Known allergy or intolerance to therapeutic agents to be tested
19. Inability to voluntarily obtain informed consent from participant or guardian
20. Perceived inability to follow study procedures and comply with protocol
21. Platelet count < 40,000 k/cumm.
22. Positive PCR test for COVID -19 within 7 days prior to the baseline day 0 visit
23. Active gastrointestinal bleeding defined as hematemesis or melena with a decrease in hemoglobin more than 2 g/dl in 24 hrs. Due to gastrointestinal bleeding, or with a decrease in mean arterial BP to < 65 mmHg.

    * Positive test is exclusionary only during screening period. If a patient tests positive any time after baseline randomization, a positive PCR test for COVID-19 will be considered as a SAE.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Indiana Universtiy, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical School, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Gawrieh S, Dasarathy S, Tu W, Kamath PS, Chalasani NP, McClain CJ, Bataller R, Szabo G, Tang Q, Radaeva S, Barton B, Nagy LE, Shah VH, Sanyal AJ, Mitchell MC; AlcHepNet Investigators. Randomized trial of anakinra plus zinc vs. prednisone for severe alcohol-associated hepatitis. J Hepatol. 2024 May;80(5):684-693. doi: 10.1016/j.jhep.2024.01.031. Epub 2024 Feb 10. PMID 38342441
- [Derived] Dasarathy S, Tu W, Bellar A, Welch N, Kettler C, Tang Q, Liangpunsakul S, Gawrieh S, Radaeva S, Mitchell M; AlcHepNet. Development and evaluation of objective trial performance metrics for multisite clinical studies: Experience from the AlcHep Network. Contemp Clin Trials. 2024 Mar;138:107437. doi: 10.1016/j.cct.2024.107437. Epub 2024 Jan 11. PMID 38215876
- See also: AlcHepNet Website — http://www.alchepnet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone: Standard of care plus prednisone 40 mg orally once daily on Days 1-30 and matching placebos for Anakinra (1 syringe s.c. once daily on Days 1-14), and zinc (matched pill once daily on Days 1-90).
  Prednisone: Prednisone is indicated for numerous conditions including inflammatory disease.
  Corticosteroids, such as prednisolone, are considered standard of care in alcoholic liver disease.
Period: Treatment
Arm/Group | Prednisone | Anakinra and Zinc
Started | 73 | 74
Completed | 30 | 20
Not Completed | 43 | 54
Not completed — Adverse Event | 9 | 5
Not completed — Met Stopping Criteria | 13 | 24
Not completed — Averse Event and Met Stopping Criteria | 2 | 9
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 11 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Other | 7 | 9
Period: Follow-up
Arm/Group | Prednisone | Anakinra and Zinc
Started | 30 | 20
Completed | 24 | 16
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Prednisone: Standard of care plus prednisone 40 mg orally once daily on Days 1-30 and matching placebos for Anakinra (1 syringe s.c. once daily on Days 1-14), and zinc (matched pill once daily on Days 1-90).
  Prednisone: Prednisone is indicated for numerous conditions including inflammatory disease.
  Corticosteroids, such as prednisolone, are considered standard of care in alcoholic liver disease.
  Placebos: Matching placebo
- Total: Total of all reporting groups
Arm/Group | Prednisone | Anakinra and Zinc | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (10.5) | 44.5 (9.3) | 44.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 41 | 47 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 61 | 65 | 126
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 61 | 60 | 121
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 73 | 74 | 147

OUTCOME MEASURES:

1. Primary Outcome: Survival at 90 Days
Description: The primary analysis will be comparisons of 90-day mortality of Prednisone and Anakinra plus zinc vs Prednisone.
Time Frame: 90 days
Measure: Number; unit: percentage of participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
percentage of participants | 90 | 70

2. Secondary Outcome: To Measure the Changes in Lille Score
Description: Change in Lille score is represented as the percentage of participants who achieved a Lille score < 0.45 on day 7.
  The Lille score will be calculated using the following website: https://www.mdcalc.com/lille-model-alcoholic-hepatitis Lille score = (exp(-R))/(1 + exp(-R)) where the variables are as follows: R = 3.19 - 0.101*(age, years) + 0.147*(albumin day 0, g/L) + 0.0165* (evolution in bilirubin level, µmol/L) - 0.206*(renal insufficiency) - 0.0065*(bilirubin day 0, µmol/L) - 0.0096*(prothrombin time, sec) Renal insufficiency = 1 (if creatinine >1.3 mg/dL (115 µmol/L)) or 0 (if ≤1.3 mg/dL (115 µmol/L)) The Lille score was developed to provide early recognition of patients with severe alcoholic hepatitis not responding to corticosteroids. Lower scores indicate more improvement in response to corticosteroids. A Lille score > 0.45 predicts worse 6-month survival. A Lille score < 0.45 predicts better 6-month survival.
Time Frame: Day 7
Population: Participant numbers may vary from participant workflow module due to the data that was able to be collected at sites and timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 59 | 61
percentage of participants | 67.8 | 65.6

3. Secondary Outcome: Changes in MELD Score
Description: The Model for End-Stage Liver Disease (MELD) is a numerical scale, ranging from 6 (less ill) to 40 (gravely ill), used for liver transplant candidates age 12 and older. It gives each person a 'score' (number) based on how urgently he or she needs a liver transplant within the next three months.
Time Frame: 7, 30, and 90 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 62 | 63
scores on a scale
  Day 7 | -2.8 (2.9) | 0.2 (4.6)
  Day 30: number analyzed (Participants) | 50 | 42
  Day 30 | -6.9 (5.3) | -1.6 (8.3)
  Day 90: number analyzed (Participants) | 33 | 28
  Day 90 | -10.3 (6.1) | -8.1 (7.1)

4. Secondary Outcome: Number of Participants With AKI (Acute Kidney Injury)
Description: * Increase in creatinine of 50% above baseline over a period of 7 days
  * Increase in creatinine of 0.3 mg/dl within a period of 48 hrs
  * Onset of renal failure requiring dialysis
Time Frame: 7, 30, and 90 days
Measure: Number; unit: Participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Participants
  Day 7 | 4 | 17
  Day 30 | 6 | 20
  Day 90 | 5 | 5

5. Secondary Outcome: Development of Multi-organ Failure
Description: Defined as failure ≥2 organs
Time Frame: 7, 30, and 90 days
Measure: Number; unit: Number of Subjects
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Number of Subjects
  Day 7 | 3 | 2
  Day 30 | 1 | 4
  Day 90 | 1 | 1

6. Secondary Outcome: Development of SIRS (Systemic Inflammatory Response Syndrome)
Description: Defined as two or more abnormalities in temperature, increased heart rate, respiration, or white blood cell count with increase in SOFA score ≥2 points
Time Frame: 7, 30, and 90 days
Measure: Number; unit: Events
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Events
  Day 7 | 0 | 2
  Day 30 | 2 | 0
  Day 90 | 1 | 0

7. Secondary Outcome: Number of Transfers to ICU
Description: Recording the change of hospital word from regular floor to ICU floor as a marker for worsening illness and care escalation
Time Frame: 7, 30, and 90 days
Measure: Number; unit: Transfers
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Transfers
  Day 7 | 2 | 5
  Day 30 | 2 | 9
  Day 90 | 2 | 0

8. Secondary Outcome: Changes in Liver Function
Description: Changes in liver function were evaluated by changes in the Child Pugh Score at days 7, 30, and 90. The Child Pugh Score is a scoring system used to assess the severity of chronic liver disease. Scores range from 5 to 15, with higher scores indicating more severe disease. Points are assigned as follows:
  Hepatic encephalopathy: None = 1 point, Grade 1 and 2 = 2 points, Grade 3 and 4 = 3 points Ascites: None = 1 point, mild = 2 points, moderate to severe = 3 points Total Bilirubin: under 2 mg/dl = 1 point, 2 to 3 mg/dl = 2 points, over 3 mg/dl = 3 points Albumin: greater than 3.5g/dl = 1 point, 2.8 to 3.5g/dl = 2 points, less than 2.8g/dl = 3 points International normalised ratio (INR): under 1.7 = 1 point, 1.7 to 2.3 = 2 points, above 2.3 = 3 points
  Assigned points for each category are summed to calculate the Child Pugh Score.
Time Frame: 7, 30, and 90 days
Population: Due to lab issues and participant follow-up at certain sites, numbers analyzed differ from lab test to timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 72 | 72
score on a scale
  Day 0 | 10.3 (1.7) | 10.1 (1.4)
  Day 7: number analyzed (Participants) | 58 | 62
  Day 7 | 9.4 (1.5) | 9.7 (1.6)
  Day 30: number analyzed (Participants) | 47 | 39
  Day 30 | 8.5 (2.0) | 9.2 (2.0)
  Day 90: number analyzed (Participants) | 30 | 24
  Day 90 | 7.2 (2.0) | 8.0 (1.8)

9. Secondary Outcome: Number of Participants With Changes in Sequential Organ Failure Assessment (SOFA) Scores and Proportions Requiring Hemodynamic Support for MAP < 65 mm Hg and Lactate > 2 mmol/l, Renal Replacement Therapy or Mechanical Ventilation.
Description: The SOFA score will be calculated at the following website https://www.mdcalc.com/sequential-organ-failure-assessment-sofa-score
  Scores can be from 0 - >14 (favorable to less favorable)
Time Frame: 180 days
Measure: Number; unit: Participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Participants
  Increase in SOFA > 2 points | 3 | 3
  Need for hemodynamic support | 9 | 11
  Renal replacement therapy | 7 | 10

10. Secondary Outcome: Number of Participants With Infections
Time Frame: 180 days
Measure: Number; unit: participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
participants | 20 | 23

11. Secondary Outcome: Number of Participants With Progression of Sepsis
Description: * Life-threatening organ dysfunction caused by a dysregulated host response to infection
  * An increase in SOFA score of 2 points of more
  * Note: most participants with severe AH have 4 points based on bilirubin only
Time Frame: 180 days
Measure: Number; unit: Participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Participants
  Sepsis | 3 | 0
  Sepsis shock | 2 | 5

12. Secondary Outcome: Percentage of Participants With Renal Dysfunction
Description: Defined by a creatinine > 2 mg/dl
Time Frame: 180 days
Measure: Number; unit: Percentage of Participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Percentage of Participants | 21.9 | 47.3

13. Secondary Outcome: Number of Participants Requiring Transfer to ICU for Care, Intubation for Airway Control, Need for Ventilator Support or RRT.
Time Frame: 180 days
Measure: Number; unit: Participant counts
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Participant counts | 6 | 15

14. Secondary Outcome: Indicators of Gut Permeability
Time Frame: 180 days
Population: Zero participants analyzed, data were not collected
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Survival
Time Frame: 30 days and 180 days
Measure: Number; unit: Percentage of Participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Percentage of Participants
  Day 30 | 97 | 85
  Day 180 | 81 | 68

16. Secondary Outcome: Transplant Free Survival Rate
Time Frame: 90 Days
Measure: Number; unit: Percentage of Participants
Arm/Group | Prednisone | Anakinra and Zinc
Number analyzed (Participants) | 73 | 74
Percentage of Participants | 88 | 64

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Prednisone | Anakinra and Zinc
All-Cause Mortality (participants affected / at risk) | 12/73 | 22/74
Serious Adverse Events (participants affected / at risk) | 41/73 | 49/74
Other Adverse Events (participants affected / at risk) | 45/73 | 51/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=73) | Anakinra and Zinc (N=74)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (7)
Abdominal pain generalized (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall hematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 13 (15) | 30 (36)
Acute post hemorrhagic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Alcohol intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcoholic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alcoholic withdrawal symptoms (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anasarca (Hepatobiliary disorders) | 4 (5) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ascites (Hepatobiliary disorders) | 2 (2) | 5 (5)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Bleeding tendencies (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood in stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
C.difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic pulmonary edema (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Central line infection (Infections and infestations) | 1 (1) | 0 (0)
Chronic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Deep vein thrombosis leg (Vascular disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Detoxification (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Encephalopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Encephalopathy hepatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Encephalopathy toxic acute (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Esophageal varices hemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Evacuation of subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Fluid overload (Cardiac disorders) | 0 (0) | 1 (1)
GI bleed (Gastrointestinal disorders) | 3 (4) | 5 (6)
Gastric ulcer hemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized edema (Cardiac disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 5 (5)
Hospice care (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Hypokalemia (Renal and urinary disorders) | 0 (0) | 3 (3)
Hyponatremia (Renal and urinary disorders) | 3 (5) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Hypotonic dehydration (Vascular disorders) | 0 (0) | 1 (1)
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Ileus of colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Internal bleeding (Vascular disorders) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Liver function test increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Macrocytic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Perineal abscess (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RUQ pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Refractory shock (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Retroperitoneal hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
SIRS (Infections and infestations) | 2 (3) | 1 (1)
STEMI (Cardiac disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic arthritis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 5 (5)
Serum creatinine increased (Renal and urinary disorders) | 2 (2) | 0 (0)
Shock (Cardiac disorders) | 0 (0) | 3 (3)
Shock circulatory (Cardiac disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 2 (2)
Subdural hematoma (Nervous system disorders) | 0 (0) | 1 (2)
Substance-induced mood disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=73) | Anakinra and Zinc (N=74)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abnormal chest sounds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Accidental overdose (therapeutic agent) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute confusional state (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 8 (9)
Agitation (Nervous system disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alcohol intoxication acute (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcoholic cirrhosis of liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy (Immune system disorders) | 1 (1) | 0 (0)
Anasarca (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Ankle edema (Cardiac disorders) | 2 (2) | 0 (0)
Ankle swelling (Cardiac disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Ascites (Hepatobiliary disorders) | 5 (5) | 6 (19)
Ascites grade 2 (Hepatobiliary disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breath sounds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Cough nonproductive (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Vascular disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ecchymosis injection site (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 2 (2) | 1 (1)
Edema dependent (Cardiac disorders) | 1 (1) | 0 (0)
Edema limbs (Cardiac disorders) | 0 (0) | 1 (1)
Edema lower limb (Cardiac disorders) | 0 (0) | 1 (1)
Edema of legs (Cardiac disorders) | 2 (4) | 3 (3)
Edema of lower extremities (Cardiac disorders) | 0 (0) | 1 (1)
Edema pulmonary (Cardiac disorders) | 0 (0) | 1 (1)
Elevated liver enzyme levels (Hepatobiliary disorders) | 3 (3) | 0 (0)
Encephalopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Encephalopathy acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Encephalopathy hepatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erythematous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Esophageal varices without mention of bleeding (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 2 (2) | 2 (2)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Gas pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrocnemius equinus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Glucose abnormal (Endocrine disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hallucinations (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 3 (4)
Hepatosplenomegaly (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 2 (3)
Hyperglycemia drug-induced (Endocrine disorders) | 1 (1) | 0 (0)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypokalemia (Renal and urinary disorders) | 7 (8) | 7 (7)
Hypomagnesaemia (Renal and urinary disorders) | 1 (1) | 2 (2)
Hyponatremia (Renal and urinary disorders) | 2 (3) | 4 (4)
Hypophosphatemia (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
INR increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infusion reaction (Immune system disorders) | 1 (1) | 0 (0)
Injection site reaction (Immune system disorders) | 3 (3) | 2 (2)
Insomnia (Nervous system disorders) | 9 (9) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Klebsiella pneumoniae pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Left upper quadrant pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 8 (9) | 4 (4)
Libido decreased (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Liver scan NOS abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Loose stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Lower leg edema (Cardiac disorders) | 1 (1) | 0 (0)
Macrocytic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mental status changes (Nervous system disorders) | 0 (0) | 1 (1)
Muscle injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (7)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 1 (1) | 3 (3)
Neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Nicotine craving (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Night sweats (General disorders) | 1 (1) | 1 (1)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paracentesis (Gastrointestinal disorders) | 1 (2) | 3 (4)
Paracentesis abdominis (Surgical and medical procedures) | 0 (0) | 1 (1)
Pedal edema (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral edema (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (nonspecific) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Restless legs (Nervous system disorders) | 0 (0) | 1 (1)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Serum creatinine increased (Renal and urinary disorders) | 0 (0) | 2 (2)
Shallow breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spider angioma (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Temperature elevation (General disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombophlebitis arm superficial (Vascular disorders) | 0 (0) | 1 (1)
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Transjugular intrahepatic portosystemic shunt (Surgical and medical procedures) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Unsteady gait (Nervous system disorders) | 1 (1) | 0 (0)
Urgency urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Vasopressin decreased urine output (Renal and urinary disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
WBC decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
WBC increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT04072822/Prot_SAP_000.pdf